CLINICAL TRIAL: NCT00298519
Title: The Influence of Maternal Ethnic Group and Diet on Breast Milk Fatty Acid Content and Its Potential Effect on Development of Allergy in the Offspring.
Brief Title: Maternal Ethnic Group,Diet,Breast Milk Fatty Acid and Potential Effect Development of Allergy in the Offspring
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Dr Chong Yap Seng, MBBS, National University Hospital, Singapore
Other Study IDs: RPR/NHG/03025
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Women of different ethnic groups have different diets that may affect the fatty acid content of their breast milk. Ethnicity may also have an independent effect on breast milk composition. The differences in fatty acid content of breast milk may influence the immune tolerance of breastfed babies, and hence the development of allergy.

DETAILED DESCRIPTION:
Pregnant women with the intention of breastfeeding their babies will be recruited about 36 weeks of gestation. After informed written consent has been obtained, a standard questionnaires will be applied to determine their demographic particulars, family of atopy and environmental details. A trained research coordinator will then profile their diet using a standard validated food frequency questionnaire (FFQ).

After delivery, these mothers will be helped to initiate, establish and continue breastfeeding. Details of their deliveries and the babies' birth measurements will be documented. A breastfeeding diary and infant/child health diary will be given to the mothers to record their breastfeeding practice as well as their child's health status.

The mothers will be followed up in the hospital before discharge, at the postnatal clinic at 1 and 6 weeks, and at 3,6 and 12 months. The mother's blood (1 ml) will be taken at 1 and 6 weeks and breast milk (20 mls) will be collected at 1 week, 6 weeks, 3 months, 6 and 12 months after delivery (as long as mothers breastfeeds).The maternal serum and breast milk total lipids will be extracted and fractionated using micro-extraction and semi-preparative liquid chromatography fraction methods. The fatty acid methyl esters will be separated, using liquid chromatography and capillary electrophoresis coupled mass spectrometry, and tje n-6 and n-3 fatty acid methyl esters identified by comparison with retention times and mass charge ratio information of pure reference substances (sigma Aldrich Sweden AB,Stockholm, Sweden).

The babies of the mothers will be followed up at 1week,6 weeks,3,6,and 12 months of age. At each visit, mothers will answer standard (ISSAC)allergy questionnaires, infant feeding patterns, hygiene practice and child's growth and development parameters: height and weight.At 12 months of age, skin prick testing will performed on the child. This method of detecting atopy is less invasive and gives faster results than measuring serum IgE levels. Our skin prick test protocol follows the routine panel used in NUH's Paediatric Allergy Clinic for under 3 years old viz. Dermatophagoides pteronyssinus (dustmite), Blomia tropicalis (dustmite), cat dander, egg white, soy protein, cow's milk, histamine positive control and saline negative control. Size of wheal and /or erythema when present will be recorded.

The fatty acid analysis of human breast milk have a very low coefficient of variation of about 2% for most of the important fatty acids and therefore 300 mothers and infants will be enough for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of about 36 weeks gestation with the intention of breastfeeding their babies.

Exclusion Criteria:

* Nil

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with the intention of breastfeeding their babies
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2003-06; Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Chong Yap Seng, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore